CLINICAL TRIAL: NCT01930435
Title: A Phase II Study Monitoring Quality of Life and Correlative Biomarkers of Mucositis in Head and Neck Cancer Patients Undergoing Radiation Therapy Utilizing a Personalized Sterile Humidification Device
Brief Title: Study of Personalized Sterile Humidification Device for Mucositis in Head and Neck Cancer Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: CC# 13202
Record Dates: First submitted 2013-08-20; First posted 2013-08-29 (Estimated); Results first posted 2017-01-12 (Estimated); Last update posted 2017-08-10 (Actual); Status verified 2017-07

CONDITIONS: Head and Neck Cancer
Keywords: Quality of Life
MeSH Terms: conditions — Head and Neck Neoplasms

STUDY DESIGN:
Intervention Model Description: humidification feasibility and efficacy
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Sterile Humidification Device, MyPurMist (Experimental): Sterile Humidification Device Twice a day, 15 minutes each 12 weeks
  Interventions: Device: Sterile Humidification Device

INTERVENTIONS:
Device: Sterile Humidification Device — This is a personal humidification device. It is hand held and produces sterile warm vapor.
  Other Names: MyPurMist

SUMMARY:
This is a single arm study of the use of a personalized sterile humidification device for 12 weeks for head and neck cancer patients undergoing radiation therapy to determine if the usage of this humidification system will result in a decrease in severity in head and neck related quality of life as measured by the MDASI HN subscale following radiation therapy as compared with historical experience. In addition, we are exploring correlative measures using CRP, IL-1, IL-6, and TNF-alpha level measurements as these are directly related to mucositis and presumably related to quality of life as indicated by the patient.

DETAILED DESCRIPTION:
The patients complete MDASI at baseline, 6 weeks, and 12 weeks. The MDASI is a validated instrument that measures symptom burden and we measure a subscale (HN) as our primary endpoint. The patients are asked to use a personal humidifier daily and complete a weekly diary showing compliance with the humidifier use.

ELIGIBILITY:
Inclusion Criteria:

* Receiving a dose of radiation therapy greater than or equal to 6000 cGy to one third of the oral cavity.
* Receiving definitive or post-operative adjuvant radiotherapy.
* Receiving radiotherapy or chemoradiation.
* Of age greater than 18 years.
* Life expectancy greater than 6 months.
* Able to provide informed consent.
* Participation of patients on other clinical trial protocols permitted, if not prohibited by trial guidelines.

Exclusion Criteria:

* Undergoing induction or neoadjuvant chemotherapy prior to radiotherapy.
* Treatment with amifostine or palifermin (keratinocyte growth factor) during radiotherapy.
* High risk for poor compliance with radiotherapy, humidification, or follow-up as assessed by the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2013-07; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sue Yom, M.D., Principal Investigator — University of California, San Francisco
Locations (1):
- Helen Diller Family Comprehensive Center, UCSF, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: Yes
sharing on request to principal investigator, case by case basis

RESULTS

PARTICIPANT FLOW:
Groups:
- Sterile Humidification Device, MyPurMist: Sterile Humidification Device Twice a day, 15 minutes each 12 weeks
  Sterile Humidification Device
Period: Overall Study
Arm/Group | Sterile Humidification Device, MyPurMist
Started | 20
Completed | 20
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Sterile Humidification Device, MyPurMist
Number analyzed (Participants) | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 12
  >=65 years | 8
Age, Continuous [Mean (Full Range); unit: years] | 62.2 [35 to 76]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 15
Region of Enrollment [Number; unit: participants]
  United States | 20

OUTCOME MEASURES:

1. Primary Outcome: Mean Change in Quality of Life as Measured by the Subscale MDASI-HN Score.
Description: The MDASI-HN assesses the severity of symptoms at their worst in the last 24 hours on a 0-10 NRS, with 0 being "not present" and 10 being "as bad as you can imagine." There are 28 items in the MDASI-HN. There are 13 general inventory items, 6 general interference items, and the HN subscale adds 9 additional items assessing mucus in the mouth and throat, difficulty swallowing/chewing, choking/coughing, difficulty with voice/speech, skin pain/burning/rash, constipation, problems with tasting food, mouth/throat sores, and problems with teeth or gums. Scores for the subscales (general, interference, HN) are averaged so that a score is obtained from 0-10 for each subscale. The mean change in quality of life is calculated as the average scores at 6 weeks minus the average of the scores at baseline. Therefore a positive value represents a worsened quality of life and a negative value is an improvement in quality of life.
Time Frame: Mean value of [(MDASI-HN score at 6 weeks) - (MDASI-HN score at baseline)]
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Sterile Humidification Device, MyPurMist
Number analyzed (Participants) | 20
units on a scale | 4.3 [3.4 to 5.3]

2. Secondary Outcome: Percentage of Patients Achieving Compliance With Use of Personalized Sterile Humidification.
Description: Compliance was pre-specified in the protocol as self-reported usage of the device at a level equal to or greater than 60% of the formal recommended usage. This cut-off at 60% represented the median of the distribution of the usage of the device among all patients. The outcome measure is the percentage of participants who reported using the device at a level equal to or greater than 60% of the total prescribed usage.
Time Frame: over entire 12 weeks duration
Measure: Number; unit: percentage of participants
Arm/Group | Sterile Humidification Device, MyPurMist
Number analyzed (Participants) | 20
percentage of participants | 65

3. Secondary Outcome: Clinician Graded CTCAE-rated Mucositis Score Over 12 Weeks
Description: The maximum severity of clinician rating of mucositis observed over 12 weeks, as graded on a scale ranging from 1 (minimal mucositis) to 3 (confluent mucositis) to 5 (death) using the Common Terminology Criteria for Adverse Events v 4.0
Time Frame: over 12 weeks duration
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Sterile Humidification Device, MyPurMist
Number analyzed (Participants) | 20
units on a scale | 3 (0.75)

4. Secondary Outcome: Rate of Feeding Tube Placement Among Patients Using Personalized Sterile Humidification
Description: Feeding Tube Placement in Patients Who Use Personalized Sterile Humidification, as determined by placement of either nasogastric or gastrostomy tube. This was enumerated as the number of participants who had a feeding tube placed.
Time Frame: over 12 weeks duration
Measure: Number; unit: participants
Arm/Group | Sterile Humidification Device, MyPurMist
Number analyzed (Participants) | 20
participants | 3

5. Secondary Outcome: Rate of Hospitalization in Patients Who Use Personalized Sterile Humidification
Description: Rate of Hospitalization in Patients Who Use Personalized Sterile Humidification, determined based on admission to hospital over active study period
Time Frame: during 12 weeks duration
Measure: Number; unit: participants
Arm/Group | Sterile Humidification Device, MyPurMist
Number analyzed (Participants) | 20
participants | 5

ADVERSE EVENTS:
Arm/Group | Sterile Humidification Device, MyPurMist
Serious Adverse Events (participants affected / at risk) | 0/20
Other Adverse Events (participants affected / at risk) | 0/20

LIMITATIONS AND CAVEATS:
The primary endpoint was based on results from a prior MDASI validation study in a similar population. However, patients enrolled in this study reported a much higher level of symptoms than was recorded in this MDASI validation study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No